CLINICAL TRIAL: NCT05309187
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation, and Dose-Expansion Study of IO-202 in Combination With Pembrolizumab in Subjects With Advanced, Relapsed, or Refractory Solid Tumors
Brief Title: Dose-Escalation and Dose-Expansion Study of IO-202 and IO-202+Pembrolizumab in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune-Onc Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IO-202-CL-002
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor, Adult
Keywords: IO-202

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IO-202 Monotherapy (dose escalation) (Experimental)
  Interventions: Biological: IO-202
- IO-202 dose escalation + pembrolizumab (Experimental): Increasing dose levels of IO-202 with fixed dose of pembrolizumab
  Interventions: Biological: IO-202 + pembrolizumab combination therapy
- IO-202 + pembrolizumab combination therapy (dose expansion) (Experimental): RP2D + pembrolizumab combination therapy in solid tumor cohorts
  Interventions: Biological: RP2D of IO-202 + pembrolizumab combination therapy in multiple solid tumor types

INTERVENTIONS:
Biological: IO-202 — IO-202 given as monotherapy
  Arms: IO-202 Monotherapy (dose escalation)
Biological: IO-202 + pembrolizumab combination therapy — IO-202 and fixed dose pembrolizumab combination therapy
  Other Names: IO-202 + Keytruda combination therapy
  Arms: IO-202 dose escalation + pembrolizumab
Biological: RP2D of IO-202 + pembrolizumab combination therapy in multiple solid tumor types — Expansion cohorts of the RP2D of IO-202 and fixed dose pembrolizumab combination therapy in multiple tumor types.
  Other Names: RP2D of IO-202 + Keytruda combination therapy
  Arms: IO-202 + pembrolizumab combination therapy (dose expansion)

SUMMARY:
To assess safety and tolerability of increasing doses of IO-202 either as monotherapy or in combination with pembrolizumab in patients with advanced solid tumors, and select the recommended Phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter, dose-escalation and dose-expansion study of IO-202 in adult subjects with advanced relapsed or refractory solid tumors to study safety, tolerability, pharmacokinetic, pharmacodynamics and clinical activity of IO-202 as monotherapy or in combination with pembrolizumab and to estimate the maximum tolerated dose (MTD) or maximum administered dose (MAD), and to select the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 years old.
2. Part 1 - Dose Escalation: Subject must have any histologically or cytologically confirmed advanced or metastatic solid tumor and has received, has been intolerant to, or has been ineligible for standard systemic therapy known to confer clinical benefit.
3. Part 2 - Dose Expansion: Subject must have failed at least one available therapy for the disease under study.
4. Subject must have measurable disease per RECIST 1.1 as assessed by local clinical site.
5. Subject must have an Eastern Cooperative Oncology Group performance status of 0 or 1.

Exclusion Criteria:

1. Subject who previously received leukocyte immunoglobulin-like receptor subfamily B (LILRB) or immunoglobulin-like transcript [ILT]) targeting agents including those targeting LILRB1 (ILT2), LILRB2 (ILT4), LILRB4 (ILT3), or leukocyte-associated immunoglobulin-like receptor 1 (LAIR1).
2. Subject who received a biologic systemic anti-cancer therapy <4 weeks or 5 half-lives prior to their first day of study drug administration, or a small molecule systemic anti-cancer therapy or definitive radiotherapy <2 weeks or 5 half-lives prior to their first day of study drug administration or have not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 Grade 1 or better from any adverse events (AEs) that were due to prior cancer therapeutics.
3. Subject has symptomatic central nervous system (CNS) tumor.
4. Requires systemic corticosteroids at a dose of >10 mg prednisone or the dose equivalent of other systemic corticosteroid.
5. History of radiation pneumonitis, non-infectious pneumonitis or interstitial lung disease.
6. History of Grade ≥3 immune-related AEs with any prior immunotherapy.
7. Subjects with known hypersensitivity to any of the components of the IO-202 formulation or pembrolizumab.
8. Active known malignancy with the exception of any of the following:

   1. Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer;
   2. Low-risk prostate cancer for which observation or hormonal therapy only is indicated;
   3. Any other malignancy treated with curative intent with the last treatment completed ≥ 6 months before study initiation (with the exception of hormonal therapies when indicated).
9. Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure (CHF) or left ventricular ejection fraction (LVEF) <40% by ECHO or multi-gated acquisition (MUGA) scan ≤28 days prior to Cycle 1 Day 1 (C1D1).
10. Any of the following in the previous 6 months: myocardial infarction, congenital long QT syndrome, Torsades de pointes, clinically significant arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), and left anterior hemiblock (bifascicular block), unstable angina, coronary/peripheral artery bypass graft, symptomatic CHF (NYHA class III or IV), cerebrovascular accident, transient ischemic attack, or pulmonary embolism. Patients with asymptomatic right bundle branch block or controlled atrial fibrillation are allowed.
11. Ongoing cardiac dysrhythmias of Grade 2 or higher per NCI CTCAE, Version 5.0.
12. Active bacterial, viral, and/or fungal infection including hepatitis B (HBV), hepatitis C, human immunodeficiency virus (HIV), severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) or acquired immunodeficiency syndrome (AIDS)-related illness.
13. Subjects with any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before study entry.
14. Subject with current active treatment in another interventional therapeutic clinical study.
15. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent and serious adverse events in patients treated with IO-202 and IO-202 + pembrolizumab | From first dose of IO-202 until the end of treatment which is up to 2 years from the first treatment date
  safety and tolerability as measured by the incidence of treatment-emergent adverse events.
Dose-limiting toxicities (DLTs) with IO-202 and IO-202 + pembrolizumab | From the first dose of IO-202 and IO-202 + pembrolizumab until 21 days after 1st treatment
  DLTs as measured by the incidence during Cycle 1.
Study discontinuations due to adverse events (AEs) | From the first dose of IO-202 IO-202 and IO-202 + pembrolizumab up to 2 years from the first treatment.
  The number of study discontinuations due to AEs

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of IO-202 | From the first dose of IO-202 until Cycle 5, Day 1
  Characterize the Cmax of IO-202 by successive sampling of blood at pre-specified times
Minimum concentration of IO-202 | From the first dose of IO-202 until the last treatment which is up to 2 years from the first treatment date
  Characterize minimum concentration of IO-202 by successive sampling of blood at pre-specified time points
Immunogenicity of IO-202 and IO-202 + pembrolizumab | From the first dose until 24 months after the last treatment
  Determine the incidence/titer of anti-drug antibodies (ADAs) against IO-202 and pembrolizumab (in combination treatment)
Anti-tumor activity of IO-202 and IO-202 + pembrolizumab | From the date of first treatment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to an estimated period of 24 months
  Determine preliminary rates of response after treatment with IO-202

OTHER OUTCOMES:
Receptor occupancy in IO-202 monotherapy and IO-202 + pembrolizumab | From the first dose of IO-202 till 21 days after
  To assess target engagement via determining Leukocyte Immunoglobulin-Like Receptor subfamily B4 (LILRB4) occupancy by IO-202 in peripheral blood myeloid cells, as expressed by % of target receptor engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Roya Nawabi, MBA, Study Director — Immune-Onc Therapeutics
Locations (10):
- United States (10):
  - USC-Norris Comprehensive Cancer Center (119), Los Angeles, California
  - University of Florida (125), Gainesville, Florida
  - Northwestern University - Feinberg School of Medicine (133), Chicago, Illinois
  - Indiana University (123), Indianapolis, Indiana
  - Tisch Mount Sinai (124), New York, New York
  - Carolina BioOncology (102), Huntsville, North Carolina
  - Sarah Cannon Research Institute/Tennessee Oncology (122), Nashville, Tennessee
  - Mary Crowley Cancer Research (108), Dallas, Texas
  - MD Anderson Cancer Center (101), Houston, Texas
  - NEXT Oncology Virginia (121), Fairfax, Virginia